CLINICAL TRIAL: NCT01280097
Title: Sleep Disruption and ICU Delirium: Delirium Assessment and Monitoring Combined With the Evaluation of Sleep Using the Sedline Brain Function Monitor.
Brief Title: Study of Sleep and Delirium in the Intensive Care Unit (ICU)
Acronym: SID
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Masimo Labs (Other)
Responsible Party: Sponsor
Other Study IDs: 10-02079
Record Dates: First submitted 2011-01-18; First posted 2011-01-20 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Delirium; Sleep Disorders, Circadian Rhythm
Keywords: Intensive care unit delirium; Sleep disruption; Sleep hygiene; Early mobilization in the Intensive care unit; Sedative agents and sleep; Circadian rhythm; Cognitive disorder; Electroencephalography (EEG) to measure sleep; Confusion Assessment Method in the Intensive Care Unit; Immune function; REM sleep
MeSH Terms: conditions — Delirium; Sleep Disorders, Circadian Rhythm; Sleep Hygiene; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected as part of the study. It will be used to measure circadian markers that will include core body temperature, cortisol and melatonin rhythms. If subjects agree, some will be stored in a bank for future research.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prospective cohort study: Observational only

SUMMARY:
The investigators will perform a prospective, cohort study of 100 older intensive care unit (ICU) patients, to investigate the association between sleep disruption and ICU delirium.

DETAILED DESCRIPTION:
Delirium and sleep disruption are both common in the intensive care unit (ICU). Delirium is a state of acute confusion, experienced especially by older adults admitted to the hospital, with the potential to adversely impact patients' outcome. Of hospitalized patients, the highest rate of delirium occurs in elderly patients in the ICU. Development of ICU delirium is associated with longer ICU and hospital length of stay, significantly higher risk of functional decline, loss of independent living, and increased mortality. Previous studies have focused on describing the clinical manifestations, risk factors and outcomes of ICU delirium; yet, the contribution of sleep timing, as well as its quality and quantity, to the development of delirium, has not previously been rigorously investigated. Sleep disturbance, including changes in sleep patterns and architecture, and decreased quality of sleep are commonly observed in older subjects. In the ICU, environmental factors (such as noise levels and continuous ambient light) and health care practices (such as frequent performance of medical procedures and tests) further contribute to sleep disruption in the critically ill older patients. Additionally, many sedative and analgesic agents potently suppress slow wave sleep. In preliminary data acquired from ICU patients, the investigators have observed that fragmented sleep is prevalent due to frequent arousals and awakenings, and that sleep architecture is altered with an increase in light sleep, and a decrease in restorative slow wave sleep. Despite the common occurrence of both ICU delirium and sleep disruption, it is not known whether sleep disruption increases the risk of developing delirium in the critically ill older patients. In this exploratory study, the investigators propose to test the hypothesis that the severity and duration of sleep disruption is an independent predictor of the onset and duration of ICU delirium in a cohort of older ICU patients. The investigators will measure sleep disruption using continuous processed electroencephalography and measure ICU delirium using a well-validated and reliable standardized instrument. Results from this study will inform the contribution of sleep disruption in the development of ICU delirium in the older critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 45 years of age admitted to the ICU, and remain for at least 24 hours.

Exclusion Criteria:

* status post craniotomy,
* moribund state with planned withdrawal of life support,
* severe dementia,
* substantial hearing impairment or inability to understand English.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include elderly patients admitted to the intensive care unit at UCSF.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2010-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
ICU delirium | Daily measurement during study
  ICU delirium will be measured using the CAM-ICU. This measurement will be done twice daily.

SECONDARY OUTCOMES:
Intensive Care Unit (ICU) length of stay | Assessed at discharge from ICU
  The day of admission to the ICU until the day of discharge from the ICU.
Hospital Length of Stay | Assesses at discharge from hospital
  This is the persons length of stay in the hospital, from admission date until discharge date.
ICU mortality | Assessed at discharge from ICU
  We will collect data on mortality during the stay in the Intensive Care Unit
Hospital mortality | Assessed at discharge from hospital
  We will assess the mortality during the hospital stay.
One year mortality | Assessed at 1 year from admission to hospital
  We will assess mortality at one year from hospital admission.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline M Leung, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States